CLINICAL TRIAL: NCT01382407
Title: Does Acne Rash During Adolescence Predict Skin Reaction to Cetuximab?
Brief Title: Does Acne Rash During Adolescence Predict Skin Reaction to Cetuximab
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: B427CTIL
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Colorectal Cancer Metastatic
Keywords: skin rash reaction; ERBITUX® (cetuximab); acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Cetuximab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cetuximab: All patients who started treatment with ERBITUX® (cetuximab), as a single agent or in combination with chemotherapy.
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab — Once a week:Loading dose-400 mg/m2;subsequent-250 mg/m2 on days 8,15, 22,29,36 if administered as a single agent, or together with Irinotecan 125 mg/m2 on days 1,8,15,29 followed by administration every 42 days.
  Other Names: Erbitux

SUMMARY:
The hypothesis of this study is that patients who suffered from acne vulgaris during adolescence are at greater risk of developing acneiform skin rash due to cetuximab.

DETAILED DESCRIPTION:
The hypothesis of this study is that patients who suffered from acne vulgaris during adolescence are at greater risk of developing acneiform skin rash due to cetuximab

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years.
* Histology or cytology proven KRAS-WT mCRC.
* Performance status ≤3 (Eastern Cooperative Oncology Group [ECOG] classification)
* Life expectancy of more than 12 weeks.
* Written informed consent.
* In women of childbearing potential, appropriate contraceptive measures must be used during treatment with cetuximab and for 6 months following the last dose of cetuximab.

Exclusion Criteria:

* Past systemic immune therapy for disease other than cancer.
* Past immune or other target therapy for cancer (not including bevacizumab).
* Presence of acne or acneiform rash prior to starting treatment with cetuximab.
* Patients with treatment plan of cetuximab and capecitabine combination.
* For female patients: the patient is pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients above the age of 18 years, who have been diagnosed with confirmed KRAS-WT mCRC, and are starting treatment with cetuximab, will be informed of the study.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-07; Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Relationship between acne and skin rash | Within Erbitux treatment period (upto 12 months)
  To determine whether there is a relationship between acne during adolescence and skin rash during cetuximab treatment?

CONTACTS AND LOCATIONS:
Overall Officials: Gil Bar-Sela, M.D., Principal Investigator — Rambam Health Care Campus
Locations (2):
- Israel (2):
  - Oncology Institute, Rambam Health Care Campus, Haifa
  - Rambam Health Care Campus, Haifa